CLINICAL TRIAL: NCT04467203
Title: A Single Center, Randomized, Open-label, Two-period Crossover Phase 1b Study to Evaluate the Effect of Food on the Pharmacokinetics of Single Oral Fadanafil Tablet in Healthy Subjects
Brief Title: Evaluate the Effects of Food on the Pharmacokinetics of Fadanafil in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5849-CPK-1002
Record Dates: First submitted 2020-06-30; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fadanafil fast to fat meal (Experimental): Seven subjects in group A will receive treatment in the following order:
  At Day 1, a single dose of Fadanafil 100mg will be administered orally after overnight fasting-> At Day 8, a single dose of Fadanafil 100mg will be administered orally with high fat meal
  Interventions: Drug: Fadanafil
- Fadanfil fat meal to fat (Experimental): Seven subjects in group B will receive treatment in the following order:
  At Day1, a single dose of Fadanafil 100mg will be administered orally with high fat meal-> At Day 8, a single dose of Fadanafil 100mg will be administered orally after overnight fasting
  Interventions: Drug: Fadanafil

INTERVENTIONS:
Drug: Fadanafil — Seven subjects in group A will receive treatment in the following order:
  At Day 1, a single dose of Fadanafil 100mg will be administered orally after overnight fasting->
  At Day 8, a single dose of Fadanafil 100mg will be administered orally with high fat meal;Seven subjects in group B will receive treatment in the following order:
  At Day1, a single dose of Fadanafil 100mg will be administered orally with high fat meal-> At Day 8, a single dose of Fadanafil 100mg will be administered orally after overnight fasting

SUMMARY:
The purpose of this study is to evaluate the effect of high fat meal on the pharmacokinetics of single oral fadanafil tablet 100mg in healthy subjects.

Fadanafil is a selective phosphodiesterase (PDE5) inhibitor. The proposed Phase 1b trial is a single center, randomized, open-label, two-period crossover study in approximately 14 Chinese healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18-45 years old, inclusive.
* Body weight ≥50kg and Body Mass Index: 19.0~26.0 kg/m2, inclusive
* The vital signs (body temperature, systolic and diastolic blood pressure, heart rate and respiration) were in the normal range, and the normal value range of each vital sign was: (1) body temperature (underarm) 36.3 ~ 37.2 ℃; (2) 90mmHg ≤ systolic blood pressure < 140mmHg; (3) 60mmhg ≤ diastolic blood pressure < 90mmHg; (4) 50th / min ≤ heart rate ≤ 90th / min.
* Before the test, a comprehensive physical examination, laboratory examination and other auxiliary examinations were carried out, and the results were normal or abnormal but of no clinical significance. The ECG QTcF < 450 ms.
* Subjects should be willing to take appropriate contraceptive measures during the period of taking the study drug and within 6 months after discontinuation to avoid pregnancy of their partners.
* Subjects understand and will comply with the study procedure, participated voluntarily and signed the informed consent.

Exclusion Criteria:

* Subjects who have a history of clinical significant drug allergy (especially those who are known or suspected to have a history of allergy to any PDE-5 inhibitor or its components) or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis) or severe allergic constitution.
* History of clinically significant ECG abnormality or family history of long QT syndrome (grandparents, parents, brothers and sisters).
* Subjects with severe systemic diseases, such as respiratory, blood, endocrine, cardiovascular and cerebrovascular diseases or mental disorders.
* Subjects with concominant diseases that may affect drug absorption, distribution, metabolism, excretion and safety evaluation, or reduce compliance.
* The test results of human immunodeficiency virus (HIV) antibody or hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody or syphilis are positive.
* Subjects who have used over-the-counter drugs, health products, Chinese herbal medicine or traditional Chinese medicine within 2 weeks before screening, or who are taking foods that affect CYP3A4, such as grapefruit or drinks containing grapefruit (except those who occasionally take paracetamol orally, but the total maximum dose cannot exceed 1g, and the drug is not allowed to take orally within 48 hours prio to first dose).
* Subjects who had used any prescription drugs (especially CYP3A4 inhibitors, nitrates, α receptor blockers, drugs potential to cause QT interval prolongation, etc.) within 4 weeks before screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter AUC(0-24) | Pre dose and 0.25, 0.5, 0.75, 1,1.5,2,2.5,4,6,8,12,24,36 hours
  AUC(0-24) of Fadanafile is area usder the curve

SECONDARY OUTCOMES:
Electrocardiogram (ECG) QT interval Safety and tolerability | Change from Baseline to 1, 2, 4, 6, 8, 12, 24 hours
  To evaluate subject ECG QT interval Changing information

CONTACTS AND LOCATIONS:
Locations (1):
- Haiyan Li, Beijing, Beijing Municipality, China